CLINICAL TRIAL: NCT04934124
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ITI 333 in Healthy Volunteers
Brief Title: Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ITI 333 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ITI-333-001; 1UG3DA047699-01 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Sequential ascending doses. Parallel (active, placebo) within each cohort
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 0.03 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 2: 0.09 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 3: 0.25 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 4: 0.75 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 5: 2.25 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 6: 6.75 mg ITI-333 or placebo (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo

INTERVENTIONS:
Drug: ITI-333 — ITI-333 oral solution
Other: Placebo — Matching placebo

SUMMARY:
The study will be conducted as a single-center, randomized, double-blind, placebo-controlled, ascending dose study in up to 8 sequential cohorts of healthy subjects. Each cohort will enroll 8 subjects: 6 subjects will receive ITI-333 and 2 subjects will receive placebo as a single oral dose after a fast of at least 10 hours.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female subjects between 18 and 45 years old (inclusive);
* BMI inclusive of 18-32 kg/m2 at screening and a minimum weight of 50 kg;
* Willingness to remain in the clinic for the inpatient portion of the study and return for follow-up visit(s) as required by protocol and as deemed necessary by the Investigator;

Key Exclusion Criteria:

* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the subject at risk or interfere with study outcome variables; this includes, but is not limited to, history of or current cardiac, hepatic, renal, neurologic, GI, pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy;
* Clinically significant abnormal findings in vital sign assessments, including blood oxygen saturation (SAO2) < 96% and < 12 breaths per min; History of psychiatric condition that in the Investigator's opinion may be detrimental to participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | up to 30 days after last dose
Change from baseline in systolic and diastolic blood pressure | Up to Day 12
Change from baseline in SAO2 | Up to Day 12
Change from baseline in ECG QT interval | Up to Day 12
Change from baseline in hemoglobin | Up to Day 12
Change from baseline in white blood cell count | Up to Day 12
Change from baseline in aspartate aminotransferase | Up to Day 12
Change from baseline in alanine aminotransferase | Up to Day 12

SECONDARY OUTCOMES:
Pharmacokinetics: AUC0-t | predose and multiple timepoints up to 96 hours postdose
  Area under the plasma concentration time curve from time zero to the last measurable of concentration of ITI-333 and metabolites
Pharmacokinetics: AUC0-inf | predose and multiple timepoints up to 96 hours postdose
  Area under the plasma concentration (ITI-333 and metabolites) time curve from time zero to infinity
Pharmacokinetics: Cmax | predose and multiple timepoints up to 96 hours postdose
  Maximum plasma concentration of ITI-333 and metabolites
Pharmacokinetics: Tmax | predose and multiple timepoints up to 96 hours postdose
  Time of maximum concentration of ITI-333 and metabolites in plasma
Pharmacokinetics: T1/2 | predose and multiple timepoints up to 96 hours postdose
  Terminal elimination half-life of ITI-333 and metabolites
Pharmacokinetics: CL/F | predose and multiple timepoints up to 96 hours postdose
  Apparent oral clearance of ITI-333
Pharmacokinetics: Vz/F | predose and multiple timepoints up to 96 hours postdose
  Apparent volume of distribution of ITI-333

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No